CLINICAL TRIAL: NCT01786525
Title: House Calls and Web-based Decision Support: Improving Access to Live Donor Kidney Transplantation
Brief Title: House Calls and Decision Support: Improving Access to Live Donor Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Rodrigue, Associate Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2012P000332; R01DK098727 (NIH)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
Keywords: Live Donor Kidney Transplantation; LDKT; African American; Disparity; Education; Patient Support
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — House Calls

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- House Calls only (Experimental): 60-minute educational intervention in patient's home which will be delivered by a health educator.
  Interventions: Behavioral: House Calls
- House Calls + Web-Based Decision Support (Active Comparator): Home based intervention plus web-based patient-centered decision support program that will be offered to participants following the home based intervention.
  Interventions: Behavioral: House Calls; Behavioral: Web-Based Patient-Centered Decision Support Intervention
- Control (No Intervention): 100 patients on the Organ Transplant Tracking Record who are not receiving the study intervention

INTERVENTIONS:
Behavioral: House Calls — 60-minute home based educational intervention which will be administered by a health educator
  Arms: House Calls + Web-Based Decision Support; House Calls only
Behavioral: Web-Based Patient-Centered Decision Support Intervention — Patients will be provided with access to the study website which will allow them to learn and receive LDKT support in a way the best meets their personal values and preferences
  Arms: House Calls + Web-Based Decision Support

SUMMARY:
The main purpose of this research program is to reduce the burden of end-stage organ disease on individuals, families, healthcare systems, and society by increasing the availability of donor organs for transplantation. Consistent with this aim, the project further examines strategies to increase access to and reduce disparities - racial, economic, gender - in live donor kidney transplantation (LDKT). Specifically, we expand the research and intensity of an innovative House Calls intervention developed by the principal investigator by including other minorities and socioeconomically disadvantaged patients and by adding a novel Patient-Centered Decision Support component. The main study hypothesis is that participants receiving the novel intervention (House Calls + Patient-Centered Decision Support) will have a higher proportion of LDKT's by the 2-year study endpoint.

DETAILED DESCRIPTION:
For most adults in late Chronic Kidney Disease (CKD Stage 4 or 5), kidney transplantation yields superior outcomes compared to long-term dialysis. Unfortunately, the demand for kidney transplantation far exceeds the supply of deceased donor organs. For those patients with healthy and willing living kidney donors, live donor kidney transplantation (LDKT) produces superior graft and patient survival rates, lower acute rejection rates, more rapid improvements in functional status, and lower healthcare costs. However, there are profound racial and income disparities in access to LDKT. Minorities, especially Blacks and Hispanics, are substantially less likely to receive LDKT compared to Whites. Also, the overall decline in LDKTs in the United States in recent years has been more pronounced for Blacks and patients with less household income. These lower LDKT rates contribute to longer waiting times for transplantation, more dialysis exposure, higher likelihood of death before transplantation, declining functional capacity, less optimal graft outcomes after transplantation, and higher healthcare costs. Therefore, interventions that expand access to LDKT, especially those targeting minority and low-income populations, are needed given the current and projected shortage of deceased donor organs.

There are several hypothesized barriers to LDKT for minorities and low-income patients, including perceived discrimination, health care mistrust, social network differences, higher rates of conditions that preclude living kidney donation, higher indirect costs of living donation, less knowledge and more concerns about LDKT, and failure to provide culturally competent education to patients and their support systems. In the last decade, the PI has developed and evaluated an innovative House Calls intervention designed to remove LDKT barriers.28-30 Health educators deliver a comprehensive and interactive program on kidney transplantation and living donation in the patient's home with members of their social network present. Relative to standard clinic-based educational programs, the House Calls intervention is superior at improving LDKT knowledge, reducing LDKT concerns, increasing LDKT willingness, and increasing rates of LDKT, particularly in minority and low-income patients (see Preliminary Studies section). However, the effectiveness of the House Calls intervention may be limited by the absence of decision-making aids, exposure to appropriate peer models, and assistance in developing an LDKT action plan beyond the House Calls intervention. This limitation and feedback from study participants have informed our strategy to enhance the House Calls intervention by incorporating a Patient-Centered Decision Support component. Additionally, there is a pressing need to identify factors that are most critical to the success of the House Calls intervention and to determine whether it can reduce the gender disparity in living kidney donation.8 Therefore, in the proposed study, we plan to pursue two primary aims and one exploratory aim:

Primary Aims

1. Evaluate the differential benefit of adding a patient-centered decision support component to the House Calls intervention. In a randomized controlled trial, we will compare House Calls (HC) alone to House Calls + Decision Support (HC+DS) in a sample of minorities and low-income patients. It is hypothesized that, compared to HC alone, the HC+DS group will have a higher proportion of patients with LDKT by the 2-yr study endpoint (primary outcome) and higher proportions of patients with ≥1 live donor inquiry, ≥1 live donor evaluation, and in LDKT Readiness Stages 4/5 by the 12-wk assessment (secondary outcomes).
2. Identify mediators of the relationship between the interventions and the occurrence of LDKT. We will investigate a set of mediators through which House Calls may increase the occurrence of LDKT, including increased LDKT knowledge, change in LDKT readiness, reduced LDKT concerns, reduced health care mistrust, the amount of time discussing LDKT with others and the quality of those interactions, and improvement in self-efficacy discussing LDKT with others.

   Exploratory Aim
3. Examine whether the House Calls intervention reduces the gender disparity in rates of living kidney donation. Women comprise 60% of all living kidney donors in the past decade. We have shown that the House Calls intervention directly educates significantly more potential living donors, including men, compared to standard clinic-based educational approaches. We hypothesize that a higher proportion of patients receiving the House Calls intervention (either HC alone or HC+DS) will have at least one potential male donor evaluated and be more likely to receive a LDKT from a male living donor, relative to a non-intervention control group, controlling for patient race/ethnicity, gender, age, and household income.

ELIGIBILITY:
Inclusion Criteria:

* non-White race/Hispanic ethnicity/low-income (250% below federal poverty guidelines)
* CKD/ESRD
* meets eligibility criteria for kidney transplant waiting list
* 21 years old or older
* self-reports being in LDKT Readiness Stage I, II, or III
* Resides within 3 hours driving time from transplant center

Exclusion Criteria:

* Awaiting combined kidney-liver transplant
* Awaiting simultaneous pancreas-kidney transplant
* Know or suspected cognitive impairment
* Prior participation in House Calls intervention study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-06; Primary Completion 2019-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this study is the proportion of enrolled patients with live donor kidney transplants | 2 years

SECONDARY OUTCOMES:
Higher proportion of enrolled patients with live donor inquires and evaluations; higher proportion of patients will be in LDKT Readiness stages 4/5 by the 12-week assessment. | 2 years

OTHER OUTCOMES:
Improvement in LDKT knowledge and LKDT readiness, reduced LDKT concerns and health care mistrust, greater amount of time spent discussing LDKT and higher quality interactions, and improvement in self-efficacy discussing LDKT. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James R Rodrigue, PhD, Principal Investigator — Beth Israel Deaconess Medical Center; Didier Mandelbrot, MD, Study Chair — Beth Israel Deaconess Medical Center; Martha Pavlakis, MS, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No